CLINICAL TRIAL: NCT00116805
Title: A Randomized, Double-Blind, Controlled Evaluation of Tenofovir DF Versus Adefovir Dipivoxil for the Treatment of HBeAg Positive Chronic Hepatitis B
Brief Title: A Study to Compare Tenofovir Disoproxil Fumarate Versus Adefovir Dipivoxil for the Treatment of HBeAg-Positive Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-174-0103; 2004-005120-41 (EudraCT Number)
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Results first posted 2010-05-19 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Chronic Hepatitis B
Keywords: tenofovir; adefovir; hepatitis B; HBeAg Positive
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Tenofovir; adefovir dipivoxil; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TDF-TDF (Experimental): TDF plus ADV placebo (double-blind period), followed by TDF (open-label period). Participants may add FTC (as part of emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) FDC tablet) to their treatment regimen in the open-label period.
  Interventions: Drug: TDF; Drug: ADV placebo; Drug: FTC/TDF
- ADV-TDF (Active Comparator): ADV plus TDF placebo (double-blind period), followed by TDF (open-label period). Participants may add FTC (as part of FTC/TDF FDC tablet) to their treatment regimen in the open-label period.
  Interventions: Drug: TDF; Drug: ADV; Drug: TDF placebo; Drug: FTC/TDF

INTERVENTIONS:
Drug: TDF — 300 mg tablet administered orally once daily
  Other Names: Viread®
Drug: ADV — 10 mg tablet administered orally once daily
  Other Names: Hepsera®
  Arms: ADV-TDF
Drug: TDF placebo — Tablet administered orally once daily
  Arms: ADV-TDF
Drug: ADV placebo — Tablet administered orally once daily
  Arms: TDF-TDF
Drug: FTC/TDF — 200/300 mg fixed-dose combination (FDC) tablet administered orally once daily
  Other Names: Truvada®

SUMMARY:
The primary objectives of this study are to compare the efficacy, safety, and tolerability of tenofovir disoproxil fumarate (TDF) versus adefovir dipivoxil (ADV) for the treatment of HBeAg-positive chronic hepatitis B. Participants will receive TDF or ADV for 48 weeks (double-blind). After 48 weeks, eligible participants switched to open-label TDF for up to 480 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible for participation in this study:

* Chronic hepatitis B virus (HBV) infection, defined as positive serum hepatitis B s-antigen (HBsAg) for more than 6 months
* 18 through 69 years of age, inclusive
* Active hepatitis B e-antigen (HBeAg) positive chronic HBV infection, with all of the following:

  * HBeAg positive at screening
  * Alanine aminotransferase (ALT) levels > 2 × ULN and ≤ 10 × the upper limit of the normal range (ULN)
  * Serum HBV DNA > 1 million copies/mL at screening
  * creatinine clearance ≥ 70 mL/min
  * hemoglobin ≥ 8 g/dL
  * neutrophils ≥ 1,000 /mL
* Knodell necroinflammatory score ≥ 3 and a Knodell fibrosis score < 4; however, up to 96 patients with cirrhosis, ie, a Knodell fibrosis score equal to 4, will be eligible for enrollment
* Negative serum β-human chorionic gonadotropin (hCG)
* Nucleotide naïve, ie, no prior nucleotide (TDF or ADV) therapy for > 12 weeks
* Nucleoside naïve, ie, no prior nucleoside (any nucleoside) therapy for > 12 weeks
* Willing and able to provide written informed consent
* Liver biopsy performed within 6 months of baseline and has readable biopsy slides or agrees to have a biopsy performed prior to baseline

Key Exclusion Criteria:

A patient who meets any of the following exclusion criteria is not to be enrolled in this study:

* Pregnant women, women who are breast feeding or who believe they may wish to become pregnant during the course of the study
* Males and females of reproductive potential who are unwilling to use an effective method of contraception during the study; for males, condoms should be used and for females, a barrier contraception method should be used
* Decompensated liver disease defined as conjugated bilirubin > 1.5 x ULN, prothrombin time (PT) > 1.5 x ULN, platelets < 75,000/mL, serum albumin < 3.0 g/dL, or prior history of clinical hepatic decompensation (eg, ascites, jaundice, encephalopathy, variceal hemorrhage)
* Received any nucleoside, nucleotide (TDF or ADV) or interferon (pegylated or not) therapy within 6 months prior to the pre-treatment biopsy
* Evidence of hepatocellular carcinoma (HCC), ie, α-fetoprotein >50 ng/mL
* Coinfection with hepatitis C virus (HCV), human immunodeficiency virus (HIV), or hepatitis delta virus (HDV)
* Significant renal, cardiovascular, pulmonary, or neurological disease
* Received solid organ or bone marrow transplantation
* Is currently receiving therapy with immunomodulators (eg, corticosteroids, etc.), investigational agents, nephrotoxic agents, or agents susceptible of modifying renal excretion
* Has proximal tubulopathy

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (78):
- United States (17):
  - Orange, California
  - Pasadena, California
  - San Diego, California
  - San Jose, California
  - Miami, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - St Louis, Missouri
  - Flushing, New York
  - New York, New York
  - Fairfax, Virginia
  - Falls Church, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Australia (10):
  - Camperdown, New South Wales
  - Concord, New South Wales
  - Westmead, New South Wales
  - Woolloongabba, Queensland
  - Clayton, Victoria
  - Footscray, Victoria
  - Parkville, Victoria
  - Prahran, Victoria
  - Fitzroy
  - Perth
- Bulgaria (2):
  - Sofia
  - Varna
- Canada (4):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnepeg, Manitoba
  - Toronto, Ontario
- Czechia (4):
  - Brno
  - Hradec Králové
  - Prague
  - Praha 6- Stresovice
- France (7):
  - Clichy
  - Grenoble
  - Lille
  - Lyon
  - Nancy
  - Paris
  - Strasbourg
- Germany (11):
  - Berlin
  - Düsseldorf
  - Essen
  - Hamburg
  - Hanover
  - Herne
  - Homburg/Saar
  - Kiel
  - Mainz
  - München
  - Tübingen
- Greece (2):
  - Athens
  - Thessaloniki
- Bologna, Italy
- Rotterdam, Netherlands
- New Zealand (4):
  - Auckland
  - Hamilton
  - Wellington
  - Whakatane
- Poland (7):
  - Bialystok
  - Bydgoszcz
  - Chorzów
  - Kielce
  - Krakow
  - Warsaw
  - Wroclaw
- Spain (2):
  - Barcelona
  - Valencia
- Turkey (Türkiye) (4):
  - Ankara
  - Bursa
  - Istanbul
  - Izmir
- United Kingdom (2):
  - Birmingham
  - London

REFERENCES:
- [Result] Kitrinos KM, Corsa A, Liu Y, Flaherty J, Snow-Lampart A, Marcellin P, Borroto-Esoda K, Miller MD. No detectable resistance to tenofovir disoproxil fumarate after 6 years of therapy in patients with chronic hepatitis B. Hepatology. 2014 Feb;59(2):434-42. doi: 10.1002/hep.26686. PMID 23939953
- [Result] Marcellin P, Gane E, Buti M, Afdhal N, Sievert W, Jacobson IM, Washington MK, Germanidis G, Flaherty JF, Aguilar Schall R, Bornstein JD, Kitrinos KM, Subramanian GM, McHutchison JG, Heathcote EJ. Regression of cirrhosis during treatment with tenofovir disoproxil fumarate for chronic hepatitis B: a 5-year open-label follow-up study. Lancet. 2013 Feb 9;381(9865):468-75. doi: 10.1016/S0140-6736(12)61425-1. Epub 2012 Dec 10. PMID 23234725
- [Result] Gordon SC, Krastev Z, Horban A, Petersen J, Sperl J, Dinh P, Martins EB, Yee LJ, Flaherty JF, Kitrinos KM, Rustgi VK, Marcellin P. Efficacy of tenofovir disoproxil fumarate at 240 weeks in patients with chronic hepatitis B with high baseline viral load. Hepatology. 2013 Aug;58(2):505-13. doi: 10.1002/hep.26277. Epub 2013 May 3. PMID 23364953
- [Result] Tsai NC, Marcellin P, Buti M, Washington MK, Lee SS, Chan S, Trinh H, Flaherty JF, Kitrinos KM, Dinh P, Charuworn P, Subramanian GM, Gane E. Viral suppression and cirrhosis regression with tenofovir disoproxil fumarate in Asians with chronic hepatitis B. Dig Dis Sci. 2015 Jan;60(1):260-8. doi: 10.1007/s10620-014-3336-7. Epub 2014 Sep 2. PMID 25179493
- [Result] Fung S, Gordon SC, Krastev Z, Horban A, Petersen J, Sperl J, Gane E, Jacobson IM, Yee LJ, Dinh P, Martins EB, Flaherty JF, Kitrinos KM, Dusheiko G, Trinh H, Flisiak R, Rustgi VK, Buti M, Marcellin P. Tenofovir disoproxil fumarate in Asian or Pacific Islander chronic hepatitis B patients with high viral load (>/= 9 log10 copies/ml). Liver Int. 2015 Feb;35(2):422-8. doi: 10.1111/liv.12694. Epub 2014 Oct 28. PMID 25277773
- [Result] Marcellin P, Buti M, Krastev Z, de Man RA, Zeuzem S, Lou L, Gaggar A, Flaherty JF, Massetto B, Lin L, Dinh P, Subramanian GM, McHutchison JG, Flisiak R, Gurel S, Dusheiko GM, Heathcote EJ. Kinetics of hepatitis B surface antigen loss in patients with HBeAg-positive chronic hepatitis B treated with tenofovir disoproxil fumarate. J Hepatol. 2014 Dec;61(6):1228-37. doi: 10.1016/j.jhep.2014.07.019. Epub 2014 Jul 18. PMID 25046847
- [Result] Buti M, Fung S, Gane E, Afdhal NH, Flisiak R, Gurel S, Flaherty JF, Martins EB, Yee LJ, Dinh P, Bornstein JD, Mani Subramanian G, Janssen HL, George J, Marcellin P. Long-term clinical outcomes in cirrhotic chronic hepatitis B patients treated with tenofovir disoproxil fumarate for up to 5 years. Hepatol Int. 2015 Apr;9(2):243-50. doi: 10.1007/s12072-015-9614-4. Epub 2015 Mar 13. PMID 25788199
- [Result] Buti M, Tsai N, Petersen J, Flisiak R, Gurel S, Krastev Z, Aguilar Schall R, Flaherty JF, Martins EB, Charuworn P, Kitrinos KM, Subramanian GM, Gane E, Marcellin P. Seven-year efficacy and safety of treatment with tenofovir disoproxil fumarate for chronic hepatitis B virus infection. Dig Dis Sci. 2015 May;60(5):1457-64. doi: 10.1007/s10620-014-3486-7. Epub 2014 Dec 23. PMID 25532501
- [Result] Liu Y, Corsa AC, Buti M, Cathcart AL, Flaherty JF, Miller MD, Kitrinos KM, Marcellin P, Gane EJ. No detectable resistance to tenofovir disoproxil fumarate in HBeAg+ and HBeAg- patients with chronic hepatitis B after 8 years of treatment. J Viral Hepat. 2017 Jan;24(1):68-74. doi: 10.1111/jvh.12613. Epub 2016 Sep 23. PMID 27658343
- [Result] Corsa A, Liu Y, Flaherty JF, Marcellin P, Miller M, Kitrinos KM. No Detectable Resistance to Tenofovir Disoproxil Fumarate (TDF) in HBeAg+ and HBeAg- Patients With Chronic Hepatitis B (CHB) After Eight Years of Treatment [Abstract 1707]. The 65th Annual Meeting of the American Association for the Study of Liver Diseases: The Liver Meeting (AASLD); 2014 08-10 November; Boston MA.
- [Result] Marcellin P, Gane EJ, Flisiak R, Trinh HN, Petersen J, Gurel S, et al. Long Term Treatment with Tenofovir Disoproxil Fumarate for Chronic Hepatitis B Infection is Safe and Well Tolerated and Associated with Durable Virologic Response with no Detectable Resistance: 8 Year Results from Two Phase 3 Trials [Abstract]. 55th Annual Meeting of the American Association for the Study of Liver Diseases (AASLD); 2014 November 7-11; Boston, MA.
- [Result] Gane EJ, Marcellin P, Sievert W, Trinh HN, Shiffman ML, Washington MK, et al. Five years of Treatment with Tenofovir DF for Chronic Hepatitis B Infection in Asian Patients is Associated with Sustained Viral Suppression and Significant Regression of Histological Fibrosis and Cirrhosis [Poster Number 1429]. 62nd Annual Meeting of the American Association for the Study of Liver Diseases; 2011 November 4-8; San Francisco, California.
- [Derived] Marcellin P, Wong DK, Sievert W, Buggisch P, Petersen J, Flisiak R, Manns M, Kaita K, Krastev Z, Lee SS, Cathcart AL, Crans G, Op den Brouw M, Jump B, Gaggar A, Flaherty J, Buti M. Ten-year efficacy and safety of tenofovir disoproxil fumarate treatment for chronic hepatitis B virus infection. Liver Int. 2019 Oct;39(10):1868-1875. doi: 10.1111/liv.14155. Epub 2019 Jul 10. PMID 31136052
- [Derived] Buti M, Wong DK, Gane E, Flisiak R, Manns M, Kaita K, Janssen HLA, Op den Brouw M, Jump B, Kitrinos K, Crans G, Flaherty J, Gaggar A, Marcellin P. Safety and efficacy of stopping tenofovir disoproxil fumarate in patients with chronic hepatitis B following at least 8 years of therapy: a prespecified follow-up analysis of two randomised trials. Lancet Gastroenterol Hepatol. 2019 Apr;4(4):296-304. doi: 10.1016/S2468-1253(19)30015-9. Epub 2019 Feb 20. PMID 30795958
- [Derived] Jacobson IM, Washington MK, Buti M, Thompson A, Afdhal N, Flisiak R, Akarca US, Tchernev KG, Flaherty JF, Aguilar Schall R, Myers RP, Subramanian GM, McHutchison JG, Younossi Z, Marcellin P, Patel K. Factors Associated With Persistent Increase in Level of Alanine Aminotransferase in Patients With Chronic Hepatitis B Receiving Oral Antiviral Therapy. Clin Gastroenterol Hepatol. 2017 Jul;15(7):1087-1094.e2. doi: 10.1016/j.cgh.2017.01.032. Epub 2017 Feb 12. PMID 28215615
- [Derived] Bayliss J, Yuen L, Rosenberg G, Wong D, Littlejohn M, Jackson K, Gaggar A, Kitrinos KM, Subramanian GM, Marcellin P, Buti M, Janssen HLA, Gane E, Sozzi V, Colledge D, Hammond R, Edwards R, Locarnini S, Thompson A, Revill PA. Deep sequencing shows that HBV basal core promoter and precore variants reduce the likelihood of HBsAg loss following tenofovir disoproxil fumarate therapy in HBeAg-positive chronic hepatitis B. Gut. 2017 Nov;66(11):2013-2023. doi: 10.1136/gutjnl-2015-309300. Epub 2016 Aug 17. PMID 27534671
- [Derived] Pan CQ, Chan S, Trinh H, Yao A, Bae H, Lou L. Similar efficacy and safety of tenofovir in Asians and non-Asians with chronic hepatitis B. World J Gastroenterol. 2015 May 14;21(18):5524-31. doi: 10.3748/wjg.v21.i18.5524. PMID 25987775
- [Derived] Heathcote EJ, Marcellin P, Buti M, Gane E, De Man RA, Krastev Z, Germanidis G, Lee SS, Flisiak R, Kaita K, Manns M, Kotzev I, Tchernev K, Buggisch P, Weilert F, Kurdas OO, Shiffman ML, Trinh H, Gurel S, Snow-Lampart A, Borroto-Esoda K, Mondou E, Anderson J, Sorbel J, Rousseau F. Three-year efficacy and safety of tenofovir disoproxil fumarate treatment for chronic hepatitis B. Gastroenterology. 2011 Jan;140(1):132-43. doi: 10.1053/j.gastro.2010.10.011. Epub 2010 Oct 16. PMID 20955704
- [Derived] Marcellin P, Heathcote EJ, Buti M, Gane E, de Man RA, Krastev Z, Germanidis G, Lee SS, Flisiak R, Kaita K, Manns M, Kotzev I, Tchernev K, Buggisch P, Weilert F, Kurdas OO, Shiffman ML, Trinh H, Washington MK, Sorbel J, Anderson J, Snow-Lampart A, Mondou E, Quinn J, Rousseau F. Tenofovir disoproxil fumarate versus adefovir dipivoxil for chronic hepatitis B. N Engl J Med. 2008 Dec 4;359(23):2442-55. doi: 10.1056/NEJMoa0802878. PMID 19052126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Australia/New Zealand. The first participant was screened on 09 June 2005. The last study visit occurred on 28 January 2016.
Pre-assignment Details: 603 participants were screened.
Groups:
- TDF-TDF: Tenofovir disoproxil fumarate (TDF) 300 mg plus placebo to match adefovir dipivoxil (ADV) (double-blind period), followed by TDF 300 mg (open-label period). Participants may have added emtricitabine (FTC) to their treatment regimen (as part of FTC 200 mg/TDF 300 mg fixed-dose combination (FDC) tablet) in the open-label period.
- ADV-TDF: ADV 10 mg plus placebo to match TDF (double-blind period), followed by TDF 300 mg (open-label period). Participants may have added FTC to their treatment regimen (as part of FTC 200 mg/TDF 300 mg FDC tablet) in the open-label period.
Period: Double-blind Period Through Week 48
Arm/Group | TDF-TDF | ADV-TDF
Started | 176 | 90
Completed | 165 | 85
Not Completed | 11 | 5
Not completed — Lost to Follow-up | 6 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrew Consent | 4 | 2
Period: Open-label Period Weeks 49 - 96
Arm/Group | TDF-TDF | ADV-TDF
Started | 154 (11 participants completed 48 weeks but did not continue on study.) | 84 (1 participant completed 48 weeks but did not continue on study.)
Completed | 144 | 83
Not Completed | 10 | 1
Not completed — Investigator's Discretion | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Safety, Tolerability, or Efficacy Reason | 1 | 0
Not completed — Seroconversion | 2 | 0
Not completed — Withdrew Consent | 2 | 1
Period: Open-label Period Weeks 97 - 144
Arm/Group | TDF-TDF | ADV-TDF
Started | 144 | 83
Completed | 133 | 74
Not Completed | 11 | 9
Not completed — Completed Study | 1 | 0
Not completed — Investigator's Discretion | 2 | 0
Not completed — Lost to Follow-up | 5 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Seroconversion | 2 | 3
Not completed — Withdrew Consent | 1 | 3
Period: Open-label Period Weeks 145 - 192
Arm/Group | TDF-TDF | ADV-TDF
Started | 133 | 74
Completed | 123 | 68
Not Completed | 10 | 6
Not completed — Completed Study | 1 | 1
Not completed — Investigator's Discretion | 2 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Safety, Tolerability, or Efficacy Reason | 0 | 1
Not completed — Seroconversion | 0 | 1
Not completed — Withdrew Consent | 3 | 2
Period: Open-label Period Weeks 193 - 240
Arm/Group | TDF-TDF | ADV-TDF
Started | 123 | 68
Completed | 110 | 64
Not Completed | 13 | 4
Not completed — Completed Study | 0 | 1
Not completed — Investigator's Discretion | 1 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Safety, Tolerability, or Efficacy Reason | 2 | 2
Not completed — Withdrew Consent | 7 | 1
Period: Open-label Period Weeks 241 - 288
Arm/Group | TDF-TDF | ADV-TDF
Started | 110 | 64
Completed | 104 | 64
Not Completed | 6 | 0
Not completed — Safety, Tolerability, or Efficacy Reason | 2 | 0
Not completed — Withdrew Consent | 4 | 0
Period: Open-label Period Weeks 289 - 336
Arm/Group | TDF-TDF | ADV-TDF
Started | 104 | 64
Completed | 98 | 57
Not Completed | 6 | 7
Not completed — Completed Study | 0 | 1
Not completed — Investigator's Discretion | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Safety, Tolerability, or Efficacy Reason | 0 | 1
Not completed — Study Site Discontinued | 0 | 1
Not completed — Withdrew Consent | 2 | 0
Period: Open-label Period Weeks 337 - 384
Arm/Group | TDF-TDF | ADV-TDF
Started | 98 | 57
Completed | 90 | 56
Not Completed | 8 | 1
Not completed — Completed Study | 1 | 0
Not completed — Investigator's Discretion | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrew Consent | 3 | 1
Period: Open-label Period Weeks 385 - 432
Arm/Group | TDF-TDF | ADV-TDF
Started | 59 (31 participants completed 384 weeks but did not continue on study.) | 30 (26 participants completed 384 weeks but did not continue on study.)
Completed | 57 | 30
Not Completed | 2 | 0
Not completed — Investigator's Discretion | 1 | 0
Not completed — Withdrew Consent | 1 | 0
Period: Open-label Period Weeks 433 - 480
Arm/Group | TDF-TDF | ADV-TDF
Started | 57 | 29 (1 participant completed 432 weeks but did not continue on study.)
Completed | 53 | 29
Not Completed | 4 | 0
Not completed — Investigator's Discretion | 1 | 0
Not completed — Withdrew Consent | 3 | 0

BASELINE CHARACTERISTICS:
Population: Randomized and Treated Analysis Set: all participants who were randomized and received at least one dose of study medication.
Groups:
- TDF-TDF: TDF 300 mg plus placebo to match ADV (double-blind period), followed by TDF 300 mg (open-label period). Participants may have added emtricitabine (FTC) to their treatment regimen (as part of FTC 200 mg/TDF 300 mg FDC tablet) in the open-label period.
- Total: Total of all reporting groups
Arm/Group | TDF-TDF | ADV-TDF | Total
Number analyzed (Participants) | 176 | 90 | 266
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 173 | 89 | 262
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11.3) | 34 (12.2) | 34 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 26 | 83
  Male | 119 | 64 | 183
Region of Enrollment [Number; unit: participants]
  United States | 30 | 14 | 44
  Greece | 1 | 2 | 3
  Spain | 7 | 2 | 9
  Turkey | 10 | 4 | 14
  Italy | 0 | 1 | 1
  United Kingdom | 6 | 1 | 7
  France | 11 | 3 | 14
  Czech Republic | 3 | 5 | 8
  Canada | 17 | 10 | 27
  Poland | 16 | 8 | 24
  Australia | 22 | 6 | 28
  Bulgaria | 17 | 11 | 28
  Germany | 20 | 8 | 28
  Netherlands | 6 | 4 | 10
  New Zealand | 10 | 11 | 21
Baseline Alanine Aminotransferase (ALT) above the Upper Limit of the Normal (ULN) Range [Number; unit: participants] — The ULN was 43 U/L for males and 34 U/L for females aged 18 to < 69, and 35 U/L for males and 32 U/L for females aged ≥ 69.
  participants
    Yes | 169 | 90 | 259
    No | 7 | 0 | 7
Prior Lamivudine or FTC Treatment [Number; unit: participants]
  Yes | 8 | 1 | 9
  No | 168 | 89 | 257
Baseline Hepatitis B Deoxyribonucleic Acid (HBV DNA) [Mean (Standard Deviation); unit: log10 copies/mL] | 8.64 (1.076) | 8.88 (0.930) | 8.72 (1.033)
Baseline Knodell Necroinflammatory Score [Mean (Standard Deviation); unit: units on a scale] — Based on Knodell numerical scoring of liver biopsy specimens. The Knodell necroinflammatory score is the combined necrosis and inflammation domain scores and ranges 0 (best) to 14 (worst).
  units on a scale | 8.3 (2.11) | 8.5 (2.07) | 8.4 (2.09)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL and Histological Improvement (2-point Reduction in Knodell Necroinflammatory Score Without Worsening in Knodell Fibrosis Score) at Week 48
Description: Complete response was a composite endpoint defined as histological response and HBV DNA < 400 copies/mL. Histological response was based on the Knodell numerical scoring of liver biopsy specimens and defined as at least a 2-point reduction in Knodell necroinflammatory score without worsening in Knodell fibrosis score. The Knodell necroinflammatory score is the combined necrosis and inflammation domain scores and ranges from 0 to 14; the Knodell fibrosis domain score ranges from 0 to 4.
  A participant was a nonresponder for the primary endpoint if either biopsy (baseline or end-of-treatment) was missing or if there was not an HBV DNA value available at or beyond Week 40.
Time Frame: Baseline; Week 48
Population: Randomized and Treated Analysis Set: all participants who were randomized and received at least one dose of study medication; the missing-equals-failure approach was used where participants with missing data were considered to have failed to reach the endpoint.
Measure: Number; unit: percentage of participants
Groups:
- TDF-TDF: TDF 300 mg plus placebo to match ADV (double-blind period), followed by TDF 300 mg (open-label period). Participants may have added FTC to their treatment regimen (as part of FTC 200 mg/TDF 300 mg FDC tablet) in the open-label period.
- ADV 10 mg: ADV 10 mg plus placebo to match TDF (double-blind period), followed by TDF 300 mg (open-label period). Participants may have added FTC to their treatment regimen (as part of FTC 200 mg/TDF 300 mg FDC tablet) in the open-label period.
Arm/Group | TDF-TDF | ADV 10 mg
Number analyzed (Participants) | 176 | 90
percentage of participants | 66.5 | 12.2
Statistical Analysis 1: Comparison: TDF-TDF vs ADV 10 mg; Test type: Non-Inferiority or Equivalence — With a sample size of 160 subjects in the TDF group and 80 subjects in the ADV group, a two group large-sample normal approximation test of proportions with a one-sided 0.025 significance level would have 95% power to reject the null hypothesis that the TDF treatment was inferior to the ADV treatment (the difference in proportions was less than -0.080) in favor of the alternative hypothesis that the TDF treatment was not inferior; p < 0.001, Z-test — P-value corresponds to a Z-test of the null hypothesis that the stratum-adjusted (baseline ALT ≤ 4 x upper limit of the normal range [ULN] or > 4 x ULN) difference is 0; 2-sided 95% confidence interval (CI), stratified by baseline ALT was used to evaluate difference between groups in proportion of complete responders; Difference in proportions = 54.1, 95% CI 2-sided [44.6 to 63.6], Standard Error of Mean 4.8

2. Secondary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL at Week 48
Time Frame: Week 48
Population: Randomized and Treated Analysis Set; the missing-equals-failure approach was used where participants with missing data were considered to have failed to reach the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 176 | 90
percentage of participants | 76.1 | 13.3
Statistical Analysis 1: Comparison: TDF-TDF vs ADV-TDF; Test type: Superiority or Other; p < 0.001, Z-test — P-value corresponds to a Z-test of the null hypothesis that the stratum-adjusted difference in zero; Difference, standard error of the difference, and the CI are stratum adjusted based on baseline ALT category (≤ 4 x ULN or > 4 x ULN); Difference in proportions = 63.1, 95% CI 2-sided [53.8 to 72.3], Standard Error of Mean 4.7

3. Secondary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL at Week 96
Time Frame: Week 96
Population: Participants in the Randomized and Treated Analysis Set with available data were analyzed. Data included for participants who discontinued study unless the discontinuation was unrelated to protocol criteria.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 165 | 86
percentage of participants | 77.6 | 77.9
Statistical Analysis 1: Comparison: TDF-TDF vs ADV-TDF; Test type: Superiority or Other; p = 0.801, Z-test — P-value corresponds to a Z-test of the null hypothesis that the stratum-adjusted difference is zero; Two-sided 95% CIs, stratified by baseline ALT (baseline ALT ≤ 4 x ULN or > 4 x ULN), were used to evaluate treatment group differences; Difference in proportions = -1.4, 95% CI 2-sided [-12.0 to 9.3], Standard Error of Mean 5.4

4. Secondary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL at Weeks 144, 192, 240, 288, 336, and 384
Time Frame: Weeks 144, 192, 240, 288, 336, and 384
Population: Randomized and Treated Analysis Set. Data included for participants who had discontinued unless the reason for discontinuation was unrelated to protocol criteria. Participants with missing values related to protocol criteria or who added FTC to their open-label TDF regimen were considered to have failed to reach the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 166 | 88
percentage of participants
  Week 144 | 71.7 | 70.5
  Week 192: number analyzed (Participants) | 165 | 88
  Week 192 | 67.9 | 71.6
  Week 240: number analyzed (Participants) | 164 | 86
  Week 240 | 63.4 | 66.3
  Week 288: number analyzed (Participants) | 163 | 88
  Week 288 | 61.3 | 64.8
  Week 336: number analyzed (Participants) | 160 | 87
  Week 336 | 59.4 | 62.1
  Week 384: number analyzed (Participants) | 155 | 86
  Week 384 | 56.1 | 60.5

5. Secondary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL at Weeks 432 and 480
Time Frame: Weeks 432 and 480
Population: Participants in the Randomized and Treated Analysis Set with observed data were analyzed; the missing-equals-excluded approach was used where participants with missing data were excluded from the analysis. Data for participants who added emtricitabine to their open-label TDF regimen were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 57 | 29
percentage of participants
  Week 432: number analyzed (Participants) | 57 | 28
  Week 432 | 93.0 | 100.0
  Week 480: number analyzed (Participants) | 51 | 29
  Week 480 | 98.0 | 96.6

6. Secondary Outcome: Change From Baseline in HBV DNA at Weeks 48, 96, 144, 192, 240, 288, 336, 384, 432, and 480
Time Frame: Baseline; Weeks 48, 96, 144, 192, 240, 288, 336, 384, 432, and 480
Population: Participants in the Randomized and Treated Analysis Set with observed data were analyzed; the missing-equals-excluded approach was used where participants with missing data were excluded from the analysis. Data for participants who added FTC to their open-label TDF regimen were included in the analysis.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 160 | 85
log10 IU/mL
  Week 48 | -6.17 (1.067) | -3.93 (1.728)
  Week 96: number analyzed (Participants) | 144 | 80
  Week 96 | -6.26 (1.137) | -6.38 (1.184)
  Week 144: number analyzed (Participants) | 131 | 72
  Week 144 | -6.32 (1.098) | -6.31 (1.407)
  Week 192: number analyzed (Participants) | 117 | 67
  Week 192 | -6.30 (1.203) | -6.49 (1.028)
  Week 240: number analyzed (Participants) | 105 | 60
  Week 240 | -6.22 (1.217) | -6.45 (0.986)
  Week 288: number analyzed (Participants) | 101 | 62
  Week 288 | -6.27 (1.248) | -6.49 (1.003)
  Week 336: number analyzed (Participants) | 94 | 57
  Week 336 | -6.35 (1.208) | -6.46 (1.017)
  Week 384: number analyzed (Participants) | 83 | 55
  Week 384 | -6.38 (1.167) | -6.28 (1.450)
  Week 432: number analyzed (Participants) | 57 | 28
  Week 432 | -6.13 (1.306) | -6.45 (1.008)
  Week 480: number analyzed (Participants) | 51 | 29
  Week 480 | -6.18 (1.300) | -6.37 (1.159)

7. Secondary Outcome: Change From Week 48 in HBV DNA at Weeks 96, 144, 192, 240, 288, 336, 384, 432, and 480
Time Frame: Week 48; Weeks 96, 144, 192, 240, 288, 336, 384, 432, and 480
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 144 | 80
log10 IU/mL
  Week 96 | -0.10 (0.422) | -2.43 (1.724)
  Week 144: number analyzed (Participants) | 131 | 72
  Week 144 | -0.19 (0.475) | -2.27 (1.866)
  Week 192: number analyzed (Participants) | 117 | 67
  Week 192 | -0.20 (0.565) | -2.41 (1.662)
  Week 240: number analyzed (Participants) | 105 | 60
  Week 240 | -0.14 (0.706) | -2.49 (1.599)
  Week 288: number analyzed (Participants) | 101 | 62
  Week 288 | -0.18 (0.762) | -2.62 (1.679)
  Week 336: number analyzed (Participants) | 94 | 57
  Week 336 | -0.25 (0.618) | -2.59 (1.622)
  Week 384: number analyzed (Participants) | 83 | 55
  Week 384 | -0.29 (0.643) | -2.34 (1.821)
  Week 432: number analyzed (Participants) | 57 | 28
  Week 432 | -0.13 (0.854) | -2.32 (1.694)
  Week 480: number analyzed (Participants) | 51 | 29
  Week 480 | -0.24 (0.630) | -2.16 (1.882)

8. Secondary Outcome: Percentage of Participants With Histological Response at Week 48
Description: Histological response was based on the Knodell numerical scoring of liver biopsy specimens and defined as at least a 2-point reduction in Knodell necroinflammatory score without worsening in Knodell fibrosis score. The Knodell necroinflammatory score is the combined necrosis and inflammation domain scores and ranges from 0 to 14; the Knodell fibrosis domain score ranges from 0 to 4.
Time Frame: Baseline; Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 176 | 90
percentage of participants
  Yes | 74.4 | 67.8
  No | 25.6 | 32.2
Statistical Analysis 1: Comparison: TDF-TDF vs ADV-TDF; Test type: Superiority or Other; p = 0.320, Z-test — P-value corresponds to a Z-test of the null hypothesis that the stratum-adjusted difference in zero. Difference, standard error of the difference, and the CI are stratum adjusted based on baseline ALT category (≤ 4 x ULN or > 4 x ULN); Difference in proportions = 5.8, 95% CI 2-sided [-5.6 to 17.2], Standard Error of Mean 5.8

9. Secondary Outcome: Percentage of Participants With Histological Response at Week 240
Description: as for outcome 8
Time Frame: Baseline; Week 240
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 76 | 48
percentage of participants
  Yes | 88.2 | 89.6
  No | 11.8 | 10.4

10. Secondary Outcome: Change From Baseline in Knodell and Ishak Necroinflammatory Scores at Week 48
Description: The Knodell necroinflammatory score is the combined score for necrosis and inflammation domains of the Knodell scoring system, and ranges from 0 (best) to 14 (worst). The Ishak score measures the degree of liver fibrosis (scarring) caused by chronic necroinflammation (inflammation leading to cell death) and ranges from 0 (best) to 6 (worst).
Time Frame: Baseline; Week 48
Population: Participants in the Randomized and Treated Analysis Set with measurements at Baseline and Week 48 were analyzed; the missing-equals-excluded approach was used where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 157 | 79
units on a scale
  Knodell Necroinflammatory Score | -3.6 (2.30) | -3.2 (2.35)
  Ishak Necroinflammatory Score | -2.7 (1.70) | -2.6 (1.94)

11. Secondary Outcome: Change From Baseline in Knodell and Ishak Necroinflammatory Scores at Week 240
Description: as for outcome 10
Time Frame: Baseline; Week 240
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 76 | 48
units on a scale
  Knodell Necroinflammatory Score | -4.8 (2.34) | -5.1 (2.43)
  Ishak Necroinflammatory Score | -4.1 (2.14) | -4.5 (2.32)

12. Secondary Outcome: Ranked Assessment of Necroinflammation and Fibrosis at Week 48
Description: Participants were ranked as having improvement, no change, worsening, or missing data (compared to Baseline) based on the Knodell scoring system, and results are presented as the percentage of participants in each category. The Knodell necroinflammatory score is the combined score for necrosis and inflammation domains of the Knodell scoring system, which ranges from 0 (best) to 14 (worst). The Knodell fibrosis domain score ranges from 0 (best) to 4 (worst). A decrease of 1 point or more indicated improvement, and an increase of 1 point or more indicated worsening.
Time Frame: Baseline; Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 176 | 90
percentage of participants
  Improvement - Necroinflammation | 81.3 | 78.9
  No Change - Necroinflammation | 4.5 | 3.3
  Worsening - Necroinflammation | 3.4 | 5.6
  Missing Data - Necroinflammation | 10.8 | 12.2
  Improvement - Fibrosis | 19.9 | 20.0
  No Change - Fibrosis | 63.6 | 61.1
  Worsening - Fibrosis | 5.1 | 6.7
  Missing Data - Fibrosis | 11.4 | 12.2

13. Secondary Outcome: Ranked Assessment of Necroinflammation and Fibrosis at Week 240
Description: as for outcome 12
Time Frame: Baseline; Week 240
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 76 | 48
percentage of participants
  Improvement - Necroinflammation | 96.1 | 97.9
  No Change - Necroinflammation | 3.9 | 2.1
  Worsening - Necroinflammation | 0 | 0
  Improvement - Fibrosis | 56.6 | 58.3
  No Change - Fibrosis | 39.5 | 39.6
  Worsening - Fibrosis | 3.9 | 2.1

14. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization at Week 48
Description: ALT normalization was defined as ALT > upper limit of normal (ULN) at baseline and within the normal range at the end of blinded treatment. The ULN was 43 U/L for males and 34 U/L for females aged 18 to < 69, and 35 U/L for males and 32 U/L for females aged ≥ 69.
Time Frame: Baseline; Week 48
Population: Participants in the Randomized and Treated Analysis Set with ALT > ULN at baseline were analyzed; the missing-equals-failure approach was used where participants with missing data were considered to have failed to reach the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 169 | 90
percentage of participants | 68.0 | 54.4
Statistical Analysis 1: Comparison: TDF-TDF vs ADV-TDF; Test type: Superiority or Other; p = 0.032, Z-test — P-value corresponds to a Z-test. Statistical tests were not adjusted for baseline ALT stratum; Difference, standard error of the difference, and CI are stratum adjusted (baseline ALT ≤ 4 x ULN or > 4 x ULN); Difference in proportions = 13.6, 95% CI 2-sided [1.1 to 26.1], Standard Error of Mean 6.4

15. Secondary Outcome: Percentage of Participants With ALT Normalization at Week 96
Description: ALT normalization was defined as ALT > ULN at baseline and within the normal range at Week 96. The ULN was 43 U/L for males and 34 U/L for females aged 18 to < 69, and 35 U/L for males and 32 U/L for females aged ≥ 69.
Time Frame: Baseline; Week 96
Population: Participants in the Randomized and Treated Analysis Set with ALT > ULN at baseline. Data included for participants who had discontinued unless the reason for discontinuation was unrelated to protocol criteria; data for participants who added FTC to their open-label TDF regimen were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 158 | 86
percentage of participants | 65.2 | 74.4
Statistical Analysis 1: Comparison: TDF-TDF vs ADV-TDF; Test type: Superiority or Other; p = 0.100, Z-test — P-value corresponds to a Z-test of the null hypothesis that the ALT stratum-adjusted difference is zero; Difference, standard error of the difference, and CI are stratum adjusted (baseline ALT ≤ 4 x ULN or > 4 x ULN); Difference in proportions = -9.8, 95% CI 2-sided [-21.5 to 1.9], Standard Error of Mean 6.0

16. Secondary Outcome: Percentage of Participants With ALT Normalization at Weeks 144, 192, 240, 288, 336, and 384
Description: ALT normalization was defined as ALT > ULN at baseline and within the normal range at the subsequent time point. The ULN was 43 U/L for males and 34 U/L for females aged 18 to < 69, and 35 U/L for males and 32 U/L for females aged ≥ 69.
Time Frame: Baseline; Weeks 144, 192, 240, 288, 336, and 384
Population: Participants in the Randomized and Treated Analysis Set with ALT > ULN at baseline and available data were analyzed. Data included for participants who had discontinued unless the reason for discontinuation was unrelated to protocol criteria; data for participants who added FTC to their open-label TDF regimen were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 161 | 87
percentage of participants
  Week 144 | 60.2 | 67.8
  Week 192: number analyzed (Participants) | 161 | 85
  Week 192 | 59.6 | 69.4
  Week 240: number analyzed (Participants) | 156 | 85
  Week 240 | 50.0 | 65.9
  Week 288: number analyzed (Participants) | 158 | 87
  Week 288 | 51.3 | 70.1
  Week 336: number analyzed (Participants) | 156 | 84
  Week 336 | 46.2 | 67.9
  Week 384: number analyzed (Participants) | 154 | 82
  Week 384 | 52.6 | 67.1

17. Secondary Outcome: Percentage of Participants With ALT Normalization at Weeks 432 and 480
Description: as for outcome 16
Time Frame: Baseline; Weeks 432 and 480
Population: Participants in the Randomized and Treated Analysis Set with ALT > ULN at baseline and with observed data were analyzed; the missing-equals-excluded approach was used where participants with missing data were excluded from the analysis. Data for participants who added FTC to their open-label TDF regimen were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 54 | 29
percentage of participants
  Week 432: number analyzed (Participants) | 54 | 28
  Week 432 | 79.6 | 78.6
  Week 480: number analyzed (Participants) | 48 | 29
  Week 480 | 75.0 | 82.8

18. Secondary Outcome: Change From Baseline in ALT at Weeks 48, 96, 144, 192, 240, 288, 336, 384, 432, and 480
Time Frame: Baseline; Weeks 48, 96, 144, 192, 240, 288, 336, 384, 432, and 480
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 160 | 84
U/L
  Week 48 | -107.2 (109.44) | -106.1 (118.90)
  Week 96: number analyzed (Participants) | 141 | 81
  Week 96 | -107.8 (108.07) | -120.4 (138.03)
  Week 144: number analyzed (Participants) | 131 | 72
  Week 144 | -100.7 (105.96) | -126.2 (150.46)
  Week 192: number analyzed (Participants) | 119 | 67
  Week 192 | -101.4 (108.63) | -139.6 (137.95)
  Week 240: number analyzed (Participants) | 102 | 62
  Week 240 | -95.9 (117.03) | -134.8 (135.59)
  Week 288: number analyzed (Participants) | 100 | 62
  Week 288 | -102.3 (111.68) | -130.9 (123.08)
  Week 336: number analyzed (Participants) | 95 | 57
  Week 336 | -101.9 (112.72) | -132.3 (125.81)
  Week 384: number analyzed (Participants) | 85 | 54
  Week 384 | -108.1 (118.05) | -133.7 (128.57)
  Week 432: number analyzed (Participants) | 57 | 28
  Week 432 | -105.0 (139.61) | -162.1 (157.83)
  Week 480: number analyzed (Participants) | 51 | 29
  Week 480 | -92.3 (83.56) | -157.5 (159.96)

19. Secondary Outcome: Change From Week 48 in ALT at Weeks 96, 144, 192, 240, 288, 336, 384, 432, and 480
Time Frame: Week 48; Weeks 96, 144, 192, 240, 288, 336, 384, 432, and 480
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 141 | 81
U/L
  Week 96 | -2.0 (17.94) | -6.9 (59.64)
  Week 144: number analyzed (Participants) | 131 | 72
  Week 144 | -0.4 (21.94) | -0.7 (82.70)
  Week 192: number analyzed (Participants) | 119 | 67
  Week 192 | -1.3 (19.57) | -7.8 (27.07)
  Week 240: number analyzed (Participants) | 102 | 62
  Week 240 | 3.7 (32.48) | -8.1 (22.92)
  Week 288: number analyzed (Participants) | 100 | 62
  Week 288 | -1.6 (19.91) | -10.3 (25.26)
  Week 336: number analyzed (Participants) | 95 | 57
  Week 336 | -1.2 (19.72) | -9.3 (22.69)
  Week 384: number analyzed (Participants) | 85 | 54
  Week 384 | -4.4 (24.87) | -6.9 (31.76)
  Week 432: number analyzed (Participants) | 57 | 28
  Week 432 | -4.3 (24.27) | -11.6 (27.09)
  Week 480: number analyzed (Participants) | 51 | 29
  Week 480 | -5.5 (19.28) | -7.1 (39.76)

20. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Loss/Seroconversion at Week 48
Description: HBeAg loss was defined as HBeAg positive at baseline and HBeAg negative at Week 48. Seroconversion to anti-HBe was defined as change of detectable antibody to HBeAg from negative at baseline to positive at Week 48.
Time Frame: Baseline; Week 48
Population: Participants in the Randomized and Treated Analysis Set who were HBeAg-positive at baseline and with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 153 | 80
percentage of participants
  HBeAg Loss | 22.2 | 17.5
  HBeAg Seroconversion | 20.9 | 17.5
Statistical Analysis 1: Comparison: TDF-TDF vs ADV-TDF; This information pertains to HBeAg loss; Test type: Superiority or Other; p = 0.245, Z-test — P-value above for HBeAg loss corresponds to a Z-test of the null hypothesis that stratum-adjusted difference is zero; Difference, standard error of the difference, and Cl are stratum adjusted based on baseline ALT category (≤ 4 x ULN or > 4 x ULN); Difference in proportions = 6.1, 95% CI 2-sided [-4.2 to 16.4], Standard Error of Mean 5.3
Statistical Analysis 2: Comparison: TDF-TDF vs ADV-TDF; This information pertains to HBeAg seroconversion; Test type: Superiority or Other; p = 0.363, Z-test — P-value for HBeAg seroconversion corresponds to Z-test of the null hypothesis that stratum-adjusted difference is zero; Difference, standard error of difference, and Cl are stratum adjusted based on baseline ALT category (≤ 4 x ULN or > 4 x ULN); Difference in proportions = 4.7, 95% CI 2-sided [-5.5 to 14.9], Standard Error of Mean 5.2

21. Secondary Outcome: Percentage of Participants With HBeAg Loss or Seroconversion to Anti-HBe at Week 96
Description: HBeAg loss was defined as HBeAg positive at baseline and HBeAg negative at Week 96. Seroconversion to anti-HBe was defined as change of detectable antibody to HBeAg from negative at baseline to positive at Week 96.
Time Frame: Baseline; Week 96
Population: Participants in the Randomized and Treated Analysis Set who were HBeAg-positive at baseline and with available data were analyzed. Data included for participants who had discontinued unless the reason for discontinuation was unrelated to protocol criteria.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 158 | 82
percentage of participants
  HBeAg Loss | 25.9 | 25.6
  Seroconversion to Anti-HBe | 22.8 | 22.0
Statistical Analysis 1: Comparison: TDF-TDF vs ADV-TDF; This information pertains to HBeAg loss; Test type: Superiority or Other; p = 0.963, Z-test — P-value above for HBeAg loss corresponds to a Z-test of the null hypothesis that stratum-adjusted difference is zero; [statistical method as in outcome 20, analysis 1]; Difference in proportions = 0.3, 95% CI 2-sided [-11.3 to 11.9], Standard Error of Mean 5.9
Statistical Analysis 2: Comparison: TDF-TDF vs ADV-TDF; This information pertains to seroconversion to anti-HBe; Test type: Superiority or Other; p = 0.904, Z-test — P-value above for HBeAg loss corresponds to a Z-test of the null hypothesis that stratum-adjusted difference is zero; Difference, standard error of the difference, and Cl are stratum adjusted based on baseline ALT category (≤ 4 x ULN or >4 x ULN); Difference in proportions = 0.7, 95% CI 2-sided [-10.4 to 11.7], Standard Error of Mean 5.6

22. Secondary Outcome: Percentage of Participants With Hepatitis B S-Antigen (HBsAg) Loss or Seroconversion at Week 48
Description: HBsAg loss was defined as HBsAg positive at baseline and HBsAg negative at Week 48. Seroconversion to anti-HBs was defined as change of detectable antibody to HBsAg from negative at baseline to positive at Week 48.
Time Frame: Baseline; Week 48
Population: Participants in the Randomized and Treated Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 158 | 82
percentage of participants
  HBsAg Loss | 3.2 | 0
  HBsAg Seroconversion | 1.3 | 0
Statistical Analysis 1: Comparison: TDF-TDF vs ADV-TDF; This information pertains to HBsAg loss; Test type: Superiority or Other; p = 0.018, Z-test — P-value corresponds to a Z-test of the null hypothesis that the ALT stratum-adjusted difference is zero. Difference, standard error of the difference, and confidence interval (CI) are stratum adjusted (baseline ALT ≤ 4 x ULN or > 4 x ULN); Difference in proportions = 10.9, 95% CI 2-sided [1.9 to 19.9], Standard Error of Mean 4.6
Statistical Analysis 2: Comparison: TDF-TDF vs ADV-TDF; This information pertains to HBsAg seroconversion; Test type: Superiority or Other; p = 0.148, Z-test — [p-value comment as in outcome 22, analysis 1]; Difference in proportions = 4.3, 95% CI 2-sided [-1.5 to 10.2], Standard Error of Mean 3.0

23. Secondary Outcome: Percentage of Participants With HBsAg Loss or Seroconversion to Anti-HBs at Week 96
Description: HBsAg loss was defined as HBsAg positive at baseline and HBsAg negative at the subsequent time point. Seroconversion to anti-HBs was defined as change of detectable antibody to HBsAg from negative at baseline to positive at the subsequent time point.
Time Frame: Baseline; Week 96
Population: Participants in the Randomized and Treated Analysis Set with available data were analyzed. Data is included for participants who had discontinued unless the reason for discontinuation was unrelated to protocol criteria.
Measure: Number; unit: percentage of participants
Groups:
- ADV-TDF: TDF 300 mg plus placebo to match ADV (double-blind period), followed by TDF 300 mg (open-label period). Participants may have added FTC to their treatment regimen (as part of FTC 200 mg/TDF 300 mg FDC tablet) in the open-label period.
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 171 | 86
percentage of participants
  HBsAg Loss | 5.3 | 5.8
  Anti-HBs Seroconversion | 4.1 | 4.7
Statistical Analysis 1: Comparison: TDF-TDF vs ADV-TDF; This information pertains to HBsAg loss; Test type: Superiority or Other; p = 0.757, Z-test — P-value above for HBsAg loss corresponds to a Z-test of the null hypothesis that stratum-adjusted difference is zero. Difference, standard error of the difference, and CI are stratum adjusted based on baseline ALT category (≤ 4 x ULN or > 4 x ULN); Difference in proportions = 0.9, 95% CI 2-sided [-4.8 to 6.5], Standard Error of Mean 2.9
Statistical Analysis 2: Comparison: TDF-TDF vs ADV-TDF; This information pertains to seroconversion to anti-HBs; Test type: Superiority or Other; p = 0.733, Z-test — P-value above corresponds to Z-test of the null hypothesis that stratum-adjusted difference is zero. Difference, standard error of the difference, and CI are stratum adjusted based on baseline ALT category (≤ 4 x ULN or > 4 x ULN); Difference in proportions = 0.9, 95% CI 2-sided [-4.2 to 5.9], Standard Error of Mean 2.6

24. Secondary Outcome: Percentage of Participants With HBsAg Loss or Seroconversion to Anti-HBs at Weeks 144, 192, 240, 288, 336, 384, 432, and 480
Description: as for outcome 23
Time Frame: Baseline; Weeks 144, 192, 240, 288, 336, 384, 432, and 480
Population: Randomized and Treated Analysis Set. Data is included for participants who had discontinued unless the reason for discontinuation was unrelated to protocol criteria. Participants with missing values related to protocol criteria or who added FTC to their open-label TDF regimen were considered to have failed to reach the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 174 | 89
percentage of participants
  HBsAg Loss - Week 144: number analyzed (Participants) | 173 | 88
  HBsAg Loss - Week 144 | 7.5 | 8.0
  Anti-HBs Seroconversion - Week 144: number analyzed (Participants) | 173 | 88
  Anti-HBs Seroconversion - Week 144 | 5.2 | 6.8
  HBsAg Loss - Week 192: number analyzed (Participants) | 171 | 89
  HBsAg Loss - Week 192 | 9.4 | 7.9
  Anti-HBs Seroconversion - Week 192: number analyzed (Participants) | 171 | 89
  Anti-HBs Seroconversion - Week 192 | 6.4 | 6.7
  HBsAg Loss - Week 240: number analyzed (Participants) | 174 | 88
  HBsAg Loss - Week 240 | 9.2 | 8.0
  Anti-HBs Seroconversion - Week 240: number analyzed (Participants) | 174 | 88
  Anti-HBs Seroconversion - Week 240 | 6.3 | 8.0
  HBsAg Loss - Week 288: number analyzed (Participants) | 173 | 88
  HBsAg Loss - Week 288 | 9.2 | 8.0
  Anti-HBs Seroconversion - Week 288: number analyzed (Participants) | 173 | 88
  Anti-HBs Seroconversion - Week 288 | 6.4 | 8.0
  HBsAg Loss - Week 336 | 10.3 | 7.9
  Anti-HBs Seroconversion - Week 336 | 7.5 | 7.9
  HBsAg Loss - Week 384: number analyzed (Participants) | 173 | 89
  HBsAg Loss - Week 384 | 11.0 | 9.0
  Anti-HBs Seroconversion - Week 384: number analyzed (Participants) | 173 | 89
  Anti-HBs Seroconversion - Week 384 | 8.1 | 7.9
  HBsAg Loss - Week 432: number analyzed (Participants) | 174 | 88
  HBsAg Loss - Week 432 | 10.9 | 10.2
  Anti-HBs Seroconversion - Week 432: number analyzed (Participants) | 172 | 87
  Anti-HBs Seroconversion - Week 432 | 7.6 | 8.0
  HBsAg Loss - Week 480 | 10.9 | 10.1
  Anti-HBs Seroconversion - Week 480 | 8.0 | 7.9

25. Secondary Outcome: Number of Participants With HBV Genotypic Changes From Baseline at Week 48 (Resistance Surveillance)
Description: Of the total number analyzed, participants evaluated for resistance included those with HBV DNA ≥ 400 copies/mL, those with viral breakthrough, and those who discontinued after Week 24 with HBV DNA ≥ 400 copies/mL.
Time Frame: Baseline; Week 48
Population: Participants in the Randomized and Treated Analysis Set were analyzed to determine if they qualified for protocol criteria for resistance surveillance, and those meeting the criteria were evaluated.
Measure: Number; unit: participants
Arm/Group | TDF-TDF | ADV-TDF
Number analyzed (Participants) | 176 | 90
participants
  Participants evaluated | 31 | 75
  Changes at conserved sites in HBV polymerase | 2 | 8
  Changes at polymorphic sites in HBV polymerase | 13 | 17
  No genotypic changes (wild-type virus) | 7 | 43
  Unable to be genotyped | 9 | 7

26. Secondary Outcome: Number of Participants With HBV Genotypic Changes From Baseline at Week 96 (Resistance Surveillance)
Description: Of the total number analyzed, participants evaluated for resistance included those with HBV DNA ≥ 400 copies/mL at Week 96 on TDF monotherapy, those with viral breakthrough, those who discontinued after Week 48 with HBV DNA ≥ 400 copies/mL, and those who added emtricitabine to the open-label TDF regimen and had HBV DNA ≥ 400 copies/mL at the time of the addition.
Time Frame: Baseline; Weeks 49 to 96
Population: Participants in the Randomized and Treated Analysis Set who continued on the study after Week 48 (ie, entered the open-label phase) were analyzed to determine if they qualified for protocol criteria for resistance surveillance, and those meeting the criteria were evaluated.
Measure: Number; unit: participants
Groups:
- TDF-TDF: TDF 300 mg plus placebo to match ADV (double-blind period), followed by TDF 300 mg (open-label period). Participants in this reporting group did not add FTC to their study regimen in the open-label period.
- TDF-TDF With Addition of FTC: TDF 300 mg plus placebo to match ADV (double-blind period), followed by TDF 300 mg (open-label period). Participants in this reporting group added FTC (as part of FTC 200 mg/TDF 300 mg FDC tablet) to their study regimen in the open-label period.
- ADV-TDF: ADV 10 mg plus placebo to match TDF (double-blind period), followed by TDF 300 mg (open-label period). Participants in this reporting group did not add FTC to their study regimen in the open-label period.
- ADV-TDF With Addition of FTC: ADV 10 mg plus placebo to match TDF (double-blind period), followed by TDF 300 mg (open-label period). Participants in this reporting group added FTC (as part of FTC 200 mg/TDF 300 mg FDC tablet) to their study regimen in the open-label period.
Arm/Group | TDF-TDF | TDF-TDF With Addition of FTC | ADV-TDF | ADV-TDF With Addition of FTC
Number analyzed (Participants) | 154 | 15 | 84 | 13
participants
  Participants evaluated | 18 | 13 | 16 | 10
  Changes at conserved sites in HBV polymerase | 2 | 0 | 2 | 3
  Changes at polymorphic sites in HBV polymerase | 3 | 1 | 1 | 2
  No genotypic changes (wild-type virus) | 10 | 5 | 12 | 3
  Unable to be genotyped | 3 | 7 | 1 | 2

27. Secondary Outcome: Number of Participants With HBV Genotypic Changes From Baseline at Week 144 (Resistance Surveillance)
Description: Of the total number analyzed, participants evaluated for resistance included those with HBV DNA ≥ 400 copies/mL at Week 144 on TDF monotherapy, those with viral breakthrough, those who discontinued after Week 96 with HBV DNA ≥ 400 copies/mL, and those who added emtricitabine to the open-label TDF regimen after Week 96 and had HBV DNA ≥ 400 copies/mL at the time of the addition.
Time Frame: Baseline; Weeks 97 to 144
Population: Participants in the Randomized and Treated Analysis Set who continued on the study after Week 96 with available data were analyzed to determine if they qualified for protocol criteria for resistance surveillance, and those meeting the criteria were evaluated.
Measure: Number; unit: participants
Arm/Group | TDF-TDF | TDF-TDF With Addition of FTC | ADV-TDF | ADV-TDF With Addition of FTC
Number analyzed (Participants) | 126 | 17 | 69 | 13
participants
  Participants evaluated | 2 | 7 | 5 | 5
  Changes at conserved sites in HBV polymerase | 1 | 2 | 2 | 0
  Changes at polymorphic sites in HBV polymerase | 0 | 3 | 3 | 0
  No genotypic changes (wild-type virus) | 1 | 2 | 0 | 3
  Unable to be genotyped | 0 | 0 | 0 | 1

28. Secondary Outcome: Number of Participants With HBV Genotypic Changes From Baseline at Week 192 (Resistance Surveillance)
Description: Of the total number analyzed, participants evaluated for resistance included those with HBV DNA ≥ 400 copies/mL at Week 192 on TDF monotherapy, those with viral breakthrough, those who discontinued after Week 144 with HBV DNA ≥ 400 copies/mL, and those who added emtricitabine to the open-label TDF regimen after Week 144 and had HBV DNA ≥ 400 copies/mL at the time of the addition.
Time Frame: Baseline; Weeks 145 to 192
Population: Participants in the Randomized and Treated Analysis Set who continued on the study after Week 144 with available data were analyzed to determine if they qualified for protocol criteria for resistance surveillance, and those meeting the criteria were evaluated.
Measure: Number; unit: participants
Arm/Group | TDF-TDF | TDF-TDF With Addition of FTC | ADV-TDF | ADV-TDF With Addition of FTC
Number analyzed (Participants) | 115 | 15 | 61 | 10
participants
  Participants evaluated | 2 | 5 | 1 | 1
  Changes at conserved sites in HBV polymerase | 0 | 0 | 0 | 0
  Changes at polymorphic sites in HBV polymerase | 1 | 0 | 1 | 1
  No genotypic changes (wild-type virus) | 0 | 1 | 0 | 0
  Unable to be genotyped | 1 | 3 | 0 | 0

29. Secondary Outcome: Number of Participants With HBV Genotypic Changes From Baseline at Week 240 (Resistance Surveillance)
Description: Of the total number analyzed, participants evaluated for resistance included those with HBV DNA ≥ 400 copies/mL at Week 240 on TDF monotherapy, those with viral breakthrough, those who discontinued after Week 192 with HBV DNA ≥ 400 copies/mL, and those who added emtricitabine to the open-label TDF regimen after Week 192 and had HBV DNA ≥ 400 copies/mL at the time of the addition.
Time Frame: Baseline; Weeks 193 to 240
Population: Participants in the Randomized and Treated Analysis Set who continued on the study after Week 192 with available data were analyzed to determine if they qualified for protocol criteria for resistance surveillance, and those meeting the criteria were evaluated.
Measure: Number; unit: participants
Arm/Group | TDF-TDF | TDF-TDF With Addition of FTC | ADV-TDF | ADV-TDF With Addition of FTC
Number analyzed (Participants) | 103 | 13 | 55 | 12
participants
  Participants evaluated | 3 | 3 | 0 | 1
  Changes at conserved sites in HBV polymerase | 0 | 0 | 0 | 1
  Changes at polymorphic sites in HBV polymerase | 2 | 0 | 0 | 0
  No genotypic changes (wild-type virus) | 1 | 2 | 0 | 0
  Unable to be genotyped | 0 | 1 | 0 | 0

30. Secondary Outcome: Number of Participants With HBV Genotypic Changes From Baseline at Week 288 (Resistance Surveillance)
Description: Of the total number analyzed, participants evaluated for resistance included those with HBV DNA ≥ 400 copies/mL at Week 288 on TDF monotherapy, those with viral breakthrough, those who discontinued after Week 240 with HBV DNA ≥ 400 copies/mL, and those who added emtricitabine to the open-label TDF regimen after Week 240 and had HBV DNA ≥ 400 copies/mL at the time of the addition.
Time Frame: Baseline; Weeks 241 to 288
Population: Participants in the Randomized and Treated Analysis Set who continued on the study after Week 240 with available data were analyzed to determine if they qualified for protocol criteria for resistance surveillance, and those meeting the criteria were evaluated.
Measure: Number; unit: participants
Arm/Group | TDF-TDF | TDF-TDF With Addition of FTC | ADV-TDF | ADV-TDF With Addition of FTC
Number analyzed (Participants) | 92 | 11 | 52 | 12
participants
  Participants evaluated | 3 | 0 | 0 | 0
  Changes at conserved sites in HBV polymerase | 0 | 0 | 0 | 0
  Changes at polymorphic sites in HBV polymerase | 0 | 0 | 0 | 0
  No genotypic changes (wild-type virus) | 2 | 0 | 0 | 0
  Unable to be genotyped | 1 | 0 | 0 | 0

31. Secondary Outcome: Number of Participants With HBV Genotypic Changes From Baseline at Week 336 (Resistance Surveillance)
Description: Of the total number analyzed, participants evaluated for resistance included those with HBV DNA ≥ 400 copies/mL at Week 336 on TDF monotherapy, those with viral breakthrough, those who discontinued after Week 288 with HBV DNA ≥ 400 copies/mL, and those who added emtricitabine to the open-label TDF regimen after Week 288 and had HBV DNA ≥ 400 copies/mL at the time of the addition.
Time Frame: Baseline; Weeks 289 to 336
Population: Participants in the Randomized and Treated Analysis Set who continued on the study after Week 288 with available data were analyzed to determine if they qualified for protocol criteria for resistance surveillance, and those meeting the criteria were evaluated.
Measure: Number; unit: participants
Arm/Group | TDF-TDF | TDF-TDF With Addition of FTC | ADV-TDF | ADV-TDF With Addition of FTC
Number analyzed (Participants) | 93 | 12 | 53 | 12
participants
  Participants evaluated | 1 | 0 | 1 | 0
  Changes at conserved sites in HBV polymerase | 0 | 0 | 0 | 0
  Changes at polymorphic sites in HBV polymerase | 0 | 0 | 0 | 0
  No genotypic changes (wild-type virus) | 0 | 0 | 1 | 0
  Unable to be genotyped | 1 | 0 | 0 | 0

32. Secondary Outcome: Number of Participants With HBV Genotypic Changes From Baseline at Week 384 (Resistance Surveillance)
Description: Of the total number analyzed, participants evaluated for resistance included those with HBV DNA ≥ 400 copies/mL at Week 384 on TDF monotherapy, those with viral breakthrough, those who discontinued after Week 336 with HBV DNA ≥ 400 copies/mL, and those who added emtricitabine to the open-label TDF regimen after Week 336 and had HBV DNA ≥ 400 copies/mL at the time of the addition.
Time Frame: Baseline; Weeks 337 to 384
Population: Participants in the Randomized and Treated Analysis Set who continued on the study after Week 336 with available data were analyzed to determine if they qualified for protocol criteria for resistance surveillance, and those meeting the criteria were evaluated.
Measure: Number; unit: participants
Arm/Group | TDF-TDF | TDF-TDF With Addition of FTC | ADV-TDF | ADV-TDF With Addition of FTC
Number analyzed (Participants) | 87 | 12 | 50 | 10
participants
  Participants evaluated | 1 | 0 | 2 | 2
  Changes at conserved sites in HBV polymerase | 0 | 0 | 1 | 0
  Changes at polymorphic sites in HBV polymerase | 0 | 0 | 1 | 1
  No genotypic changes (wild-type virus) | 0 | 0 | 0 | 1
  Unable to be genotyped | 1 | 0 | 0 | 0

33. Secondary Outcome: Number of Participants With HBV Genotypic Changes From Baseline at Week 432 (Resistance Surveillance)
Description: Of the total number analyzed, participants evaluated for resistance included those with HBV DNA ≥ 400 copies/mL at Week 432 on TDF monotherapy, those with viral breakthrough, those who discontinued after Week 384 with HBV DNA ≥ 400 copies/mL, and those who added emtricitabine to the open-label TDF regimen after Week 384 and had HBV DNA ≥ 400 copies/mL at the time of the addition.
Time Frame: Baseline; Weeks 385 to 432
Population: Participants in the Randomized and Treated Analysis Set who continued on the study after Week 384 with available data were analyzed to determine if they qualified for protocol criteria for resistance surveillance, and those meeting the criteria were evaluated.
Measure: Number; unit: participants
Arm/Group | TDF-TDF | TDF-TDF With Addition of FTC | ADV-TDF | ADV-TDF With Addition of FTC
Number analyzed (Participants) | 49 | 10 | 26 | 4
participants
  Participants evaluated | 1 | 3 | 0 | 1
  Changes at conserved sites in HBV polymerase | 0 | 0 | 0 | 0
  Changes at polymorphic sites in HBV polymerase | 1 | 0 | 0 | 0
  No genotypic changes (wild-type virus) | 0 | 3 | 0 | 1
  Unable to be genotyped | 0 | 0 | 0 | 0

34. Secondary Outcome: Number of Participants With HBV Genotypic Changes From Baseline at Week 480 (Resistance Surveillance)
Description: Of the total number analyzed, participants evaluated for resistance included those with HBV DNA ≥ 400 copies/mL at Week 480 on TDF monotherapy, those with viral breakthrough, those who discontinued after Week 432 with HBV DNA ≥ 400 copies/mL, and those who added emtricitabine to the open-label TDF regimen after Week 432 and had HBV DNA ≥ 400 copies/mL at the time of the addition.
Time Frame: Baseline; Weeks 433 to 480
Population: Participants in the Randomized and Treated Analysis Set who continued on the study after Week 432 with available data were analyzed to determine if they qualified for protocol criteria for resistance surveillance, and those meeting the criteria were evaluated.
Measure: Number; unit: participants
Arm/Group | TDF-TDF | TDF-TDF With Addition of FTC | ADV-TDF | ADV-TDF With Addition of FTC
Number analyzed (Participants) | 47 | 10 | 26 | 3
participants
  Participants evaluated | 0 | 3 | 1 | 0
  Changes at conserved sites in HBV polymerase | 0 | 0 | 0 | 0
  Changes at polymorphic sites in HBV polymerase | 0 | 1 | 0 | 0
  No genotypic changes (wild-type virus) | 0 | 2 | 1 | 0
  Unable to be genotyped | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 480
Description: Randomized and Treated Analysis Set: all participants who were randomized and received at least one dose of study drug.
Groups:
- Double-Blind TDF: Adverse events this reporting group include those occurring in the TDF-TDF group during the double-blind period only (baseline to Week 48).
  TDF 300 mg plus placebo to match ADV (double-blind period).
- Double-Blind ADV: Adverse events this reporting group include those occurring in the ADV-TDF group during the double-blind period only (baseline to Week 48).
  ADV 10 mg plus placebo to match TDF (double-blind period).
- Open-Label TDF: Adverse events for this reporting group include those occurring during the open-label TDF 300 mg period (Week 49 up to Week 480), regardless of which group they were randomized to in the double-blind period.
  TDF 300 mg + ADV placebo or ADV 10 mg + TDF placebo (double-blind period), followed by TDF 300 mg (open-label period). Participants may have added FTC to their treatment regimen (as part of FTC 200 mg/TDF 300 mg FDC tablet) in the open-label period.
Arm/Group | Double-Blind TDF | Double-Blind ADV | Open-Label TDF
Serious Adverse Events (participants affected / at risk) | 15/176 | 7/90 | 41/238
Other Adverse Events (participants affected / at risk) | 97/176 | 49/90 | 165/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind TDF (N=176) | Double-Blind ADV (N=90) | Open-Label TDF (N=238)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 1
Congenital anomaly in offspring (Congenital, familial and genetic disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 1
Abscess soft tissue (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 4 | 6
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Glucose urine present (Investigations) | 0 | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Tonsillar neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1
Facial spasm (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 2
Drug dependence (Psychiatric disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 3
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind TDF (N=176) | Double-Blind ADV (N=90) | Open-Label TDF (N=238)
Abdominal pain (Gastrointestinal disorders) | 6 | 3 | 22
Abdominal pain upper (Gastrointestinal disorders) | 15 | 4 | 25
Diarrhoea (Gastrointestinal disorders) | 12 | 3 | 12
Nausea (Gastrointestinal disorders) | 26 | 1 | 9
Fatigue (General disorders) | 22 | 8 | 20
Influenza like illness (General disorders) | 9 | 3 | 14
Seasonal allergy (Immune system disorders) | 4 | 1 | 17
Bronchitis (Infections and infestations) | 2 | 4 | 13
Influenza (Infections and infestations) | 8 | 5 | 25
Nasopharyngitis (Infections and infestations) | 22 | 13 | 43
Upper respiratory tract infection (Infections and infestations) | 7 | 6 | 21
Creatinine renal clearance decreased (Investigations) | 1 | 1 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 3 | 18
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 5 | 11
Dizziness (Nervous system disorders) | 12 | 2 | 11
Headache (Nervous system disorders) | 31 | 14 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 30
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 18
Hypertension (Vascular disorders) | 3 | 1 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and investigator may publish or present the results of the trial generated there with prior written consent of Gilead; or 2 years after the trial has ended at all institutions. Proposed publications/target venue must go to Gilead 30 days (manuscripts) or 15 days (abstracts/presentations) prior. Any Gilead confidential information in the document(s) must be deleted, or if requested publication delayed for up to 45 days to permit Gilead to obtain intellectual property protection.